CLINICAL TRIAL: NCT05920824
Title: Clinical Phenotypes, Risk Factors, & Determinants of Outcome in Functional Mitral and Tricuspid Valve Regurgitation
Brief Title: Atrial Functional Mitral Regurgitation and Tricuspid Regurgitation
Status: Recruiting | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 326447
Record Dates: First submitted 2023-06-16; First posted 2023-06-27 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation; Functional Mitral Regurgitation; Functional Tricuspid Regurgitation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Echocardiogram — Ultrasound scan of the heart

SUMMARY:
A prospective, observational cohort study designed to identify clinical phenotypes and evaluate predictors & outcomes of functional mitral and tricuspid valve regurgitation in patients with atrial fibrillation.

Participant will under go:

* Baseline echocardiography
* Cpex Echocardiography
* Blood test: BNP
* 1 year follow up Echocardiography

Participants will be stratified into three subgroups:

* Atrial Functional MR
* Atrial Functional TR
* Mixed MR & TR

DETAILED DESCRIPTION:
Rationale

The natural history and risk factors for atrial valve disease are poorly understood and characterised. This study will examine differences between atrial mitral and atrial tricuspid disease and help us understand the natural history of these pathologies.

Study objectives

Primary objective

* Identify & characterise phenotypes in functional mitral and tricuspid valve regurgitation
* Identify risk factors for progression of disease and outcome.

Secondary objective

Compare the three groups: atrial functional MR, atrial functional TR, and mixed disease, and identify any differences/similarities.

Primary endpoint

Effective Regurgitant Orifice Area at 1 year

Secondary endpoint

* Progression of valve disease defined as worsening of mitral or tricuspid regurgitation > 1 grade at 1 year.
* Functional: New York Heart Association Class, Predicted VO2max (<84%).
* Heart Failure admission within 1 year of recruitment.
* Mortality.

Recruitment will take place from the out-patient clinics & echocardiography laboratory at St Bartholomew's Hospital

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age of 18 years or older
* Atrial fibrillation
* Moderate or severe atrial valve disease
* Adequate 2D echocardiography views including parasternal long axis, short axis, apical two chamber, apical three chamber and four chamber.

Exclusion Criteria:

* Unwilling or unable to give consent
* Left ventricular impairment (ejection fraction < 50%).
* Primary/organic valve disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment will take place from the out-patient clinics & echocardiography laboratory at St Bartholomew's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 141 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Effective Regurgitant Orifice Area at 1 year | 1 year
  Measure the EROA by echocardiography after 1 year

SECONDARY OUTCOMES:
Progression of valve disease defined as worsening of mitral or tricuspid regurgitation > 1 grade at 1 year. | 1 year
  Measure the change in regurgitation severity
Functional: New York Heart Association Class, Predicted VO2max (<84%). | 1 year
  Evaluate participants' physical abilities and endurance, focusing on two key measures: The New York Heart Association (NYHA) Functional Classification and the predicted maximum oxygen uptake (VO2max)
Heart Failure admission within 1 year of recruitment. | 1 year
  incidence of heart failure admissions within a one-year period following the recruitment of participants.
Mortality | 1 year
  Document and analyze the mortality rates among participants

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev bhattacharyya, Principal Investigator — Barts & The London NHS Trust; Jawza Aldakhil, Study Chair — Barts & The London NHS Trust
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided